CLINICAL TRIAL: NCT06930794
Title: An Open-label, Randomized, Controlled, Multicenter Phase IIIb Clinical Study to Evaluate the Efficacy and Safety of Vebreltinib Enteric Capsule Combined With Platinum-based Doublet Chemotherapy Compared With Platinum-based Doublet Chemotherapy in Subjects With Locally Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer Who Have Not Received Previous Systemic Treatment and MET-Positive
Brief Title: A Study of Vebreltinib and Platinum-Containing Double Agents in Subjects With MET-Positive
Acronym: KUNPENG-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Pearl Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLB1001-IIIb-NSCLC-02
Record Dates: First submitted 2025-02-27; First posted 2025-04-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The experimental group will receive the treatment regimen of Vebreltinib combined with platinum-base (Experimental): Vebreltinib: Each cycle is 3 weeks (21 days). It is administered orally twice a day (BID), and the dosage level depends on the cohort assignment.
  Platinum-based doublet chemotherapy: Each cycle is 3 weeks (21 days), and it is administered once on the first day (D1) of each cycle. Pemetrexed at a dose of 500 mg/m² plus a platinum agent (carboplatin with an area under the curve (AUC) of 5 or cisplatin at a dose of 75 mg/m²) is given by intravenous infusion for 4 to 6 cycles as the initial treatment. After that, it is switched to pemetrexed (500 mg/m²) given by intravenous infusion as the maintenance treatment.
  Interventions: Drug: Vebreltinib combined with platinum-based doublet chemotherapy.
- The comparator group will receive the platinum-based doublet chemotherapy regimen. (Active Comparator): Platinum-based doublet chemotherapy: Each cycle is 3 weeks (21 days), and it is administered once on the first day (D1) of each cycle. Pemetrexed at a dose of 500 mg/m² plus a platinum agent (carboplatin with an area under the curve (AUC) of 5 or cisplatin at a dose of 75 mg/m²) is given by intravenous infusion for 4 to 6 cycles as the initial treatment. After that, it is switched to pemetrexed (500 mg/m²) given by intravenous infusion as the maintenance treatment.
  Interventions: Drug: platinum-based doublet chemotherapy.

INTERVENTIONS:
Drug: Vebreltinib combined with platinum-based doublet chemotherapy. — Vebreltinib: Each cycle is 3 weeks (21 days). It is administered orally twice a day (BID), and the dosage level depends on the cohort assignment.
  Platinum-based doublet chemotherapy: Each cycle is 3 weeks (21 days), and it is administered once on the first day (D1) of each cycle. Pemetrexed at a dose of 500 mg/m² plus a platinum agent (carboplatin with an area under the curve (AUC) of 5 or cisplatin at a dose of 75 mg/m²) is given by intravenous infusion for 4 to 6 cycles as the initial treatment. After that, it is switched to pemetrexed (500 mg/m²) given by intravenous infusion as the maintenance treatment.
  Arms: The experimental group will receive the treatment regimen of Vebreltinib combined with platinum-base
Drug: platinum-based doublet chemotherapy. — Platinum-based doublet chemotherapy: Each cycle is 3 weeks (21 days), and it is administered once on the first day (D1) of each cycle. Pemetrexed at a dose of 500 mg/m² plus a platinum agent (carboplatin with an area under the curve (AUC) of 5 or cisplatin at a dose of 75 mg/m²) is given by intravenous infusion for 4 to 6 cycles as the initial treatment. After that, it is switched to pemetrexed (500 mg/m²) given by intravenous infusion as the maintenance treatment.
  Arms: The comparator group will receive the platinum-based doublet chemotherapy regimen.

SUMMARY:
This study is an open-label, randomized, controlled, multicenter Phase IIIb clinical study, aiming to evaluate the efficacy, safety, and tolerability of Vebreltinib Enteric Capsule combined with platinum-based doublet chemotherapy compared with platinum-based doublet chemotherapy in treating subjects with locally advanced or metastatic non-squamous NSCLC who have not received previous systemic treatment and MET-positive.

The target population of this study is subjects with histologically confirmed locally advanced or metastatic non-squamous NSCLC who have not received previous systemic anti-tumor treatment and MET-positive( MET Amplification or Overexpression).

This study adopts an enrichment design. The enriched population is those with MET GCN ≥ 6, and the overall population is those with MET GCN ≥ 4.

This study consists of two parts: the lead-in period (Part 1) and the randomized controlled period (Part 2). Both the lead-in period (Part 1) and the randomized controlled period (Part 2) will include a screening period (from Day -28 to Day -1), a treatment period (until the termination of treatment), and a follow-up period (including safety follow-up and survival follow-up).

DETAILED DESCRIPTION:
Part 1 (Lead-in Period):

The lead-in period is set before the randomized controlled period, aiming to evaluate the safety, tolerability, and preliminary efficacy of Vebreltinib Enteric Capsule combined with platinum-based doublet chemotherapy, and to determine the recommended dose of Vebreltinib Enteric Capsule combined with platinum-based doublet chemotherapy. Initially, it is planned to set up 2 dose groups in the lead-in period. After the screening period, eligible subjects will be assigned to the 2 dose cohorts in chronological order, and the subjects will receive oral treatment of Vebreltinib Enteric Capsule at different doses combined with intravenous chemotherapy of standard-dose platinum-based doublet according to the cohort assignment.

Vebreltinib Enteric Capsule: Each cycle is 3 weeks (21 days), administered orally twice a day (BID), and the dose level depends on the cohort assignment.

Platinum-based doublet chemotherapy: Each cycle is 3 weeks (21 days), and it is administered once on Day 1 (D1) of each cycle. Pemetrexed 500 mg/m² + platinum (carboplatin AUC5 or cisplatin 75 mg/m²) is given by intravenous infusion for 4 to 6 cycles as the initial treatment, and then it is switched to pemetrexed (500 mg/m²) by intravenous infusion as the maintenance treatment.

In this part, the "3+3" dose escalation design will be adopted to determine the maximum tolerated dose (MTD) and/or the recommended dose of the combination of Vebreltinib Enteric Capsule and platinum-based doublet treatment in subjects with locally advanced or metastatic non-squamous NSCLC.

Part 2 (Randomized Controlled Period):

After completing the lead-in period study in Part 1, once the investigator and the sponsor have determined the recommended dose of the combination of Vebreltinib Enteric Capsule, the randomized controlled study in Part 2 will be carried out to evaluate the efficacy of Vebreltinib Enteric Capsule combined with platinum-based doublet chemotherapy compared with platinum-based doublet chemotherapy in subjects with locally advanced or metastatic non-squamous NSCLC carrying MET amplification.

After the screening period, eligible subjects will be stratified according to the stratification factors (baseline brain metastasis status [yes vs no], MET gene copy number [GCN] [≥4 and <6 vs ≥6 and <10 vs ≥10]) and randomly assigned to the experimental group or the control group at a 1:1 allocation ratio using the stratified block randomization method. The experimental group will receive the treatment regimen of Vebreltinib Enteric Capsule combined with platinum-based doublet chemotherapy, and the control group will receive the platinum-based doublet chemotherapy regimen.

Subjects randomly assigned to the control group will have the opportunity to choose to receive single-agent treatment with Vebreltinib Enteric Capsule (200 mg BID) after the disease progression is evaluated by the investigator and confirmed by the blinded independent central review (BICR). Receiving single-agent treatment with Vebreltinib Enteric Capsule after progression is not mandatory and is determined by the investigator at his/her own discretion (subject to the approval of the sponsor).

Number of subjects: It is expected to enroll 6-18 subjects in the dose escalation stage of the lead-in period, and about 20-40 subjects in the cohort expansion stage, with a total of about 26-58 subjects to be enrolled (the final number will depend on the number of dose levels). The planned sample size of the enriched population with GCN≥6 in the randomized controlled period is 182 cases. Considering that the proportion of the enriched population with GCN≥6 in the general population is approximately 75%, the estimated sample size of the total population is 242.

Independent Data Monitoring Committee (IDMC): During the interim analysis, the independent statistical team of the IDMC will conduct the interim analysis, which will be evaluated by the IDMC experts, and the IDMC will give its recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. male or female subjects ≥ 18 years of age at the time of signing ICF.
2. histologically or cytologically confirmed diagnosis of non-radical, locally advanced (Stage IIIB and IIIC) or metastatic (Stage IV) non-squamous cell type NSCLC (refer to the American Joint Committee on Cancer [AJCC] Lung Cancer Stages, 8th edition for lung cancer staging criteria).
3. Part 1 (introductory stage)Subjects with MET-positive (MET amplification or MET overexpression) tumors will be enrolled. MET amplification is defined as the presence of MET amplification confirmed by second-generation sequencing (NGS) or fluorescence in situ hybridization (FISH) with a mean MET GCN ≥ 4 cells/cell or MET/CEP7 ≥ 2. MET overexpression is defined as c-Met showing strong positive (3+) staining in ≥50% of tumor cells as determined by immunohistochemistry (IHC) (central laboratory results). And subjects are required to provide sufficient tumor tissue (archived or fresh samples) for retrospective analysis in the central laboratory (see Laboratory Manual) to support the development of concomitant diagnostic reagents required for the marketing of Vebreltinib. Part 2 (Randomized Control Phase) MET amplification is defined as subjects' tumor tissue (archived or fresh samples) with an average MET GCN ≥ 4 cells/cell or MET/CEP7 ≥ 2 as confirmed by fluorescence in situ hybridization (FISH) in the central laboratory, and subjects will be required to provide sufficient tumor tissue (archived or fresh samples) for retrospective assay analysis by a central laboratory (see Laboratory Manual). Laboratory Manual) to support the development of concomitant diagnostic reagents required for the marketing of Vebreltinib.
4. Part 1 (Lead-in Period): Documented evidence confirms that the tumor tissue specimen tested negative for sensitive epidermal growth factor receptor (EGFR) mutations (including exon 19 deletion, exon 21 L858R or L861Q mutations, exon 18 G719X mutations, exon 20 S768I/T790M mutations, or exon 20 insertion mutations), ALK fusion-negative, ROS1 fusion-negative, and MET exon 14 skipping mutation-negative. Additionally, if the subject has already undergone testing for BRAF V600E mutation, NTRK fusion, RET fusion, or ERBB2 (HER-2) mutation, the results must be negative.

   Part 2 (Randomized Controlled Period): Documented evidence confirms that the tumor tissue specimen tested negative for sensitive EGFR mutations (including exon 19 deletion, exon 21 L858R or L861Q mutations, exon 18 G719X mutations, exon 20 S768I/T790M mutations, or exon 20 insertion mutations), ALK fusion-negative, ROS1 fusion-negative, and MET exon 14 skipping mutation-negative. Additionally, if the subject has already undergone testing for BRAF V600E mutation, KRAS mutation, NTRK fusion, RET fusion, or ERBB2 (HER-2) mutation, the results must be negative.
5. no prior systemic therapy for locally advanced or metastatic non-squamous NSCLC. Note: Subjects are permitted to receive neoadjuvant/adjuvant therapy as long as the relevant therapy has been completed for at least 6 months prior to disease diagnosis of locally progressive or metastatic tumor.
6. at least one measurable target lesion as defined by the Response to Criteria for Evaluation of Efficacy in Solid Tumors (RECIST) V1.1 criteria (see Chapter 10.4).
7. ECOG PS ≤ 1.
8. expected survival ≥ 12 weeks as determined by the investigator.
9. good organ function as determined by medical evaluation (within 7 days prior to first study dose), including:

   * Good hematologic status, defined as absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, hemoglobin ≥ 90 g/L, platelets ≥ 100 x 10^9/L. No platelet transfusions within 3 days prior to the test, no red blood cell transfusions within 14 days prior to the test, and no hematopoietic growth factor therapy within 7 days prior to the test (polyethylene glycolated granulocyte colony-stimulating factor [G-CSF] or erythropoietin [EPO] within 14 days prior to testing).
   * Good hepatic function, defined as serum TBIL ≤ 1.5 x ULN (TBIL ≤ 3 x ULN and direct bilirubin [DBIL] ≤ 1.5 x ULN in subjects known to have Gilbert's syndrome), serum ALT/AST ≤ 2.5 x ULN (≤ 5.0 x ULN for subjects with confirmed liver metastases) .
   * The organ function is well-determined by medical evaluation (within 7 days prior to the first study drug administration), including:
   * Good renal function , defined as: creatinine clearance rate ≥50 mL/min (≥60 mL/min for those receiving cisplatin, calculated using the Cockcroft-Gault formula).
   * Good coagulation function, defined as (including when receiving anticoagulation): prothrombin time (PT) < 1.5 x ULN and activated partial thromboplastin time (APTT) < 1.5 x ULN If subjects are receiving anticoagulant therapy, they must have received a stabilized dose of anticoagulant for at least 1 month prior to the first study dose.
10. Female subjects must be using adequate contraception and not breastfeeding during study participation and for 90 days after completion of study treatment; female subjects of childbearing potential must have had a serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test performed within 7 days prior to the first dose of the drug and be negative; and female subjects of no childbearing potential must meet one of the following criteria at screening:

    * Reached postmenopausal status, refer to the NCCN Breast Cancer Guidelines (2024 V3.0) for a detailed definition of menopause.
    * Have undergone and documented irreversible sterilization such as hysterectomy, bilateral salpingo-oophorectomy, or bilateral salpingo-oophorectomy (not tubal ligation).
11. Male subjects of childbearing potential must use adequate contraception (e.g., barrier methods of contraception) during study participation and for 90 days after completion of study treatment. Male subjects must also refrain from sperm donation during study participation and for 90 days after the last dose of study treatment.
12. be able to provide a signed ICF that complies with the requirements and restrictions outlined in the ICF and this study protocol.

Exclusion Criteria:

1. has participated in another therapeutic clinical trial within 28 days prior to the first study dose.
2. have undergone major surgery within 28 days prior to the first study dose or anticipate the need for major surgery during the study period. Diagnostic procedures such as thoracoscopic biopsy and mediastinoscopy may be enrolled 7 days after the procedure. No waiting period is required after implantable infusion port and catheter placement.
3. lung field or whole brain radiotherapy within 28 days prior to first study dose or palliative localized radiotherapy within 14 days prior to first study dose.
4. have received a proprietary Chinese medicine with an antitumor indication within 1 week prior to the first study dose. Has received local antitumor drug therapy (e.g., thoracic or abdominal perfusion, etc.) within 14 days or 5 half-lives, whichever is shorter, prior to the first study dose.
5. a history of another primary malignancy diagnosed or requiring treatment within the past 3 years (with the exception of localized basal cell carcinoma of the skin or squamous cell carcinoma of the skin, which has been adequately treated, or any other carcinoma in situ currently in complete remission)
6. toxicity from prior therapy that has not returned to ≤ Grade 1 or baseline levels (as assessed by NCI-CTCAE v5.0), except for alopecia, skin pigmentation, and any other toxicity that is assessed by the investigator to be stable and does not affect the safety of participation in this study
7. presence of clinically symptomatic CNS metastases. Note: Subjects with symptomatic CNS metastases may be enrolled in the study after they have been treated and their symptoms are controlled, have no lesion progression for at least 2 weeks during the Screening Period as confirmed by clinical and imaging studies, and have not had an increase in their steroid dose (<10 mg/day of prednisolone or its equivalent) for the management of CNS symptoms in the 4 weeks prior to the first study dose.

   Those with combined carcinomatous meningitis or meningeal spread or spinal cord compression were not eligible for enrollment, regardless of whether they had clinical symptoms.
8. subjects with poorly controlled clinical third space effusions, including but not limited to pleural effusions, abdominal effusions, or pericardial effusions, who, in the judgment of the investigator, are not suitable for enrollment.
9. presence of severe cardiovascular or cerebrovascular disease, including but not limited to:

   * Mean QT interval (QTcF) corrected by the Fridericia formula from three ECG examinations at rest > 470 ms.
   * Symptomatic heart failure with a New York Heart Association (NYHA) cardiac function classification of II or higher (see Chapter 10.6).
   * Echocardiographic (ECHO) assessment showing a baseline left ventricular ejection fraction (LVEF) below the lower limit of institutional normal (LLN) or <50%.
   * Any clinically significant rhythmic, conduction, or morphologic abnormality as demonstrated by resting ECG results, such as complete left bundle branch block, third-degree heart block, and ventricular arrhythmias requiring antiarrhythmic drug therapy.
   * Presence of any factor that increases the risk of QTc prolongation or the risk of arrhythmia, such as heart failure, Severe hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or use of any comorbid medication known to prolong the QT interval within 14 days prior to the first dose of study treatment.
   * Any of the following within 6 months prior to first study administration: myocardial infarction, severe/unstable angina, coronary artery bypass grafting, congestive heart failure, cardiomyopathy, pulmonary embolism, cerebrovascular accident, or transient ischemic attack.
10. the presence of serious or uncontrolled systemic disease, as judged by the Investigator, including but not limited to:

    * Uncontrolled hypertension, defined as a systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg despite pharmacological treatment Subjects with a history of hypertension will be allowed to enroll if their blood pressure control is stable on antihypertensive therapy and within the above ranges.
    * Current unstable or clinically significant interstitial lung disease or interstitial pneumonia, or high risk of interstitial lung disease or interstitial pneumonia (e.g., interfering with activities of daily living or requiring therapeutic intervention).
    * Unstable or decompensated other systemic disease, deep vein thrombosis, active bleeding, etc.
11. presence of uncontrolled co-infections, including but not limited to:

    - Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection. If hepatitis B surface antigen (HBsAg) positive, HBV DNA testing should be performed. If the HBV DNA test value is ≤500 IU/mL (or 2000 copies/mL), the subject is eligible to participate in the study.

    If HCV antibody positive, HCV RNA testing should be performed. If HCV RNA is negative, the subject is eligible to participate in the study.
    * Known human immunodeficiency virus (HIV) infection or known history of acquired immunodeficiency syndrome (AIDS).
    * Active Syphilis positive infection.
    * Active tuberculosis infection.
    * Other active infection requiring systemic therapy within 14 days prior to the first study dose.
12. presence of dysphagia, or active gastrointestinal disease, or major gastrointestinal surgery that may interfere with the administration or absorption of Vebreltinib (e.g., refractory nausea/vomiting/diarrhea, ulcerative lesions, malabsorption syndrome, etc.).
13. hypersensitivity to Pertinib or its excipients, or history of allergic reaction to drugs with similar chemical or biological structure or analogs to Pertinib, or history of severe allergic reaction to Pemetrexed, Cisplatin, Carboplatin (NCI CTCAE v5.0 ≥ Grade 3).
14. have received any live attenuated vaccination within 30 days prior to the first study dose.
15. known psychiatric or substance abuse disorders that may affect study compliance.
16. the presence of other conditions that, in the investigator's assessment, make participation in the study inappropriate, such as participation in a study that, in the investigator's opinion, is not in the subject's best interest, or that may increase the risk of toxicity, or that may interfere with absorption, distribution, metabolism, or excretion of the study medication, or that may impair the assessment of study results, or that the subject is not able to comply with the study protocols and study limitations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Introductory phase-Dose-limiting toxicity (DLT) Incidence of DLT events during the observation period | 1 year
  laboratory tests, vital signs, physical examination, electrocardiogram (ECG), and the Eastern United States Collaborative Oncology Group (ECOG) clinically significant abnormal values in physical status (PS).To evaluated DLT events during the observation period.
Incidence and severity of adverse events (AEs) . | 1 year
  laboratory tests, vital signs, physical examination, electrocardiogram (ECG), and the Eastern United States Collaborative Oncology Group (ECOG) clinically significant abnormal values in physical status (PS).
Introductory phase-Recommended dosage for MTD and/or co-administration. | 1 year
  Confirm Recommended dosage for MTD and/or co-administration.
Randomized control period-Progression-free survival (PFS) as assessed by the Blinded Independent Center Review Board (BICR) according to RECIST V1.1 in the MET GCN ≥6-enriched population. | 4 years
  Progression Free Survival is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD or death due to any cause.
Randomized control period-Progression-free survival (PFS) as assessed by BICR according to the criteria for evaluating the efficacy of solid tumors (RECIST V1.1) in the full MET GCN ≥4 population. | 4 years
  Progression Free Survival is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD or death due to any cause.

SECONDARY OUTCOMES:
Introductory phase-Objective Response Rate (ORR) as assessed by the investigator according to RECIST V1.1. | 2 years
  Objective response rate is defined as the percentage of patients who experienced either a complete response (CR) or partial response (PR) from first administration of trial treatment to first observation of progressive disease (PD).
Introductory phase-Duration of Remission (DoR) as assessed by the investigator according to RECIST V1.1. | 2 years
  Duration of remission is defined as the time from the first tumor assessment as CR or PR to the first assessment of PD (Progressive Disease) or death from any cause.
Introductory phase-Disease control rate (DCR) as assessed by the investigator according to RECIST V1.1. | 2 years
  Disease Control Rate according to RECIST 1.1 is the percentage of patients who experienced either a complete response (CR), partial response (PR) or stable disease (SD).
Introductory phase-Progression-free survival (PFS), 6-month PFS rate as assessed by the investigator according to RECIST V1.1. | 2 years
  Progression Free Survival is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD or death due to any cause.
Introductory phase-6-month overall survival (OS) rate as assessed by the investigator according to RECIST V1.1. | 2 years
  Overall Survival is defined as the length of time from the start of treatment (or diagnosis) until death from any cause.
Introductory phase-Blood drug concentration of Vebreltinib | 1 year
  Assess the area under the plasma concentration-time curve (AUC0-t, AUC0-∞) of Vebreltinib.
Introductory phase-Blood drug concentration of Vebreltinib | 1 year
  Assess the maximum plasma concentration (Cmax) of Vebreltinib.
Introductory phase-Blood drug concentration of Vebreltinib | 1 year
  Assess the time to reach peak concentration (Tmax) of Vebreltinib.
Introductory phase-Blood drug concentration of Vebreltinib | 1 year
  Assess the elimination half-life (t½) of Vebreltinib.
Introductory phase-Blood drug concentration of Vebreltinib | 1 year
  Assess the apparent systemic clearance (CL/F) of Vebreltinib.
Introductory phase-Companion Diagnostics, CDx | 4 years
  All subjects in the study are required to provide sufficient tumor tissues (either archived or fresh samples) and blood samples for testing and analysis, in order to support the development of companion diagnostic reagents for the marketing of Vebreltinib.
  MET gene copy number in patient tumor tissue detected by FISH and in patient blood detected by NGS.
Randomized control period-PFS as assessed by the investigator according to RECIST V 1.1. | 4 years
  Progression Free Survival is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD or death due to any cause.
Randomized control period-Objective remission rate (ORR) as assessed by the investigator according to RECIST V1.1. | 4 years
  Objective response rate is defined as the percentage of patients who experienced either a complete response (CR) or partial response (PR) from first administration of trial treatment to first observation of progressive disease (PD).
Randomized control period-Disease control rate (DCR) as assessed by the investigator according to RECIST V1.1. | 4 years
  Disease Control Rate according to RECIST 1.1 is the percentage of patients who experienced either a complete response (CR), partial response (PR) or stable disease (SD).
Randomized control period-Duration of remission (DoR) as assessed by BICR and by the investigator according to RECIST V1.1. | 4 years
  Duration of remission is defined as the time from the first tumor assessment as CR or PR to the first assessment of PD (Progressive Disease) or death from any cause.
Randomized control period-Overall survival (OS) as assessed by BICR and by the investigator according to RECIST V1.1. | 4 years
  Overall Survival is defined as the length of time from the start of treatment (or diagnosis) until death from any cause.
Randomized control period-Incidence and severity of adverse events (AEs) (based on NCI-CTCAE V5.0); | 4 years
  clinically significant abnormal values seen in laboratory tests, vital signs, physical examination, electrocardiogram (ECG), and Eastern US Collaborative Oncology Group (ECOG) physical status (PS).
Randomized control period-Blood drug concentration of Vebreltinib. | 1 year
  Assess the area under the plasma concentration-time curve (AUC0-t, AUC0-∞) of Vebreltinib.
Randomized control period-Blood drug concentration of Vebreltinib. | 1 year
  Assess the maximum plasma concentration (Cmax) of Vebreltinib.
Randomized control period-Blood drug concentration of Vebreltinib. | 1 year
  Assess the time to reach peak concentration (Tmax) of Vebreltinib.
Randomized control period-Blood drug concentration of Vebreltinib. | 1 year
  Assess the elimination half-life (t½) of Vebreltinib.
Randomized control period-Blood drug concentration of Vebreltinib. | 1 year
  Assess the apparent systemic clearance (CL/F) of Vebreltinib.
Randomized control period-Companion Diagnostics, CDx | 4 years
  All subjects in the study are required to provide sufficient tumor tissues (either archived or fresh samples) and blood samples for testing and analysis, in order to support the development of companion diagnostic reagents for the marketing of Vebreltinib.
  MET gene copy number in patient tumor tissue detected by FISH and in patient blood detected by NGS.

OTHER OUTCOMES:
Introductory phase-Drug resistance related mechanism. | 4 years
  Subject is encouraged to provide blood samples (optional) at baseline and disease progression for retrospective analysis to explore mechanisms of resistance in molecular genes to Vebreltinib.
  Expression of ctDNA in patient blood detected by NGS.
Randomized control period- Second progression-free survival (PFS2) as assessed by the investigators. | 4 years
  Progression Free Survival is defined as the time (in months) from the first administration of trial treatment to the date of the first documentation of PD or death due to any cause.
Randomized control period- Subject Health-Related Quality of Life (HRQoL) assessment: European Five Dimensional Health Scale (EQ-5D-5L). | 4 years
  Health status includes 5 dimensions of mobility, self-care, daily activities, pain or discomfort, anxiety or depression. The five dimensions can be represented by the numbers 1-5. And the EQ-VAS assessment, patient can indicate health status with the numbers 0-100.
Randomized control period- To compare the differences in clinical efficacy of brentinib in combination with platinum-containing two-agent chemotherapy in different MET GCN populations. | 4 years
  To explore the correlation between MET gene copy number (GCN) and clinical efficacy of Vebreltinib.
  PFS in patients with MET GCN ≥4 or ≥6.
Randomized control period-Drug resistance related mechanism. | 4 years
  Subject is encouraged to provide blood samples (optional) at baseline and disease progression for retrospective analysis to explore mechanisms of resistance in molecular genes to Vebreltinib.
  Expression of ctDNA in patient blood detected by NGS.

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, MD, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China